CLINICAL TRIAL: NCT01514656
Title: Hospital-based CPR Training for At-risk Family Members Using a Video-self Instruction Kit or Video-only
Brief Title: CPR Training: Video Self-Instruction Kit or Video-Only
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRS- 814676
Record Dates: First submitted 2011-12-12; First posted 2012-01-23 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Cardiovascular Risk Factors; Coronary Disease; Cardiac Arrest
MeSH Terms: conditions — Coronary Disease; Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Video Self-Instruction (VSI) kit (Active Comparator): Individuals will learn CPR using American Heart Association's Video Self-Instruction kit. Main data points being collected at various increments over 12 months are: 1) CPR quality at 6 to 12 months 2) Comfort Level using the skills they learned
  Interventions: Other: CPR Training using the Family and Friends CPR Anytime Video Self Instruction
- Video-only (Experimental): Individuals will learn CPR skills using a Video training method. Main data points being collected at various increments over 12 months are: 1) CPR Skills at 6 to 12 months 2) Comfort Level with using CPR
  Interventions: Other: CPR Training using the Family and Friends CPR Anytime Video Self Instruction
- Recruitment with Volunteers (Active Comparator): Volunteer subjects will be identified by hospital stakeholders, and they will be given surveys to assess their confidence, attitudes and beliefs towards this program at 3-month integrals.
  Interventions: Other: Implementation of a Hospital-based CPR Training Model
- Recruitment with Nurses (Active Comparator): Nurse subjects will be identified by hospital stakeholders, and they will be given surveys to assess their confidence, attitudes and beliefs towards this program at 3-month integrals.
  Interventions: Other: Implementation of a Hospital-based CPR Training Model
- Prompting to practice skills (Active Comparator): Individuals will be prompted every two months and encouraged to practice the skills that they learned. Main data points being collected at various increments over 12 months are: 1) Comfort Level with using CPR 2) CPR Skills at 6 to 12 months.
  Interventions: Other: Follow-up prompting to encourage skill retention
- No prompting to practice skills (Active Comparator): Individuals will not be prompted to practice skills. Main data points being collected at various increments over 12 months are: 1) Comfort Level with using CPR 2) CPR Skills at 6 to 12 months.
  Interventions: Other: Follow-up prompting to encourage skill retention

INTERVENTIONS:
Other: CPR Training using the Family and Friends CPR Anytime Video Self Instruction — Subjects will be trained using the American Heart Association's Family and Friends CPR Anytime Program. The subject's will undergo training in-hospital then they will be encouraged to take the training materials home with them to practice CPR with their family members and friends.
  Arms: Video Self-Instruction (VSI) kit; Video-only
Other: Implementation of a Hospital-based CPR Training Model — Nurses and Volunteers will be trained in the hospital-based CPR Training Model, and be encouraged to implement the training program in their respective hospitals.
  Arms: Recruitment with Nurses; Recruitment with Volunteers
Other: Follow-up prompting to encourage skill retention — Subjects will be contacted every two months and encouraged to practice the skills that they have learned. Means of contact include: a) email b) text blasts c) phone calls d) social media e) mail
  Arms: No prompting to practice skills; Prompting to practice skills

SUMMARY:
Prompt delivery of cardiopulmonary resuscitation (CPR) is a crucial determinant of survival for many victims of sudden cardiac arrest (SCA), yet bystander CPR is provided in less than one third of witnessed SCA events. A number of barriers to bystander CPR training have been identified including time and cost of the training course. Since the large majority of arrest events occur in the home environment, studies have suggested that providing CPR training to family members of hospitalized cardiac patients may serve as a useful approach to address an environment in which bystander CPR is frequently not provided. Utilizing an existing in-hospital program to train adult family members, the investigators will assess the skills of those who learn CPR through two different education methods (video-only and video self-instruction (VSI) kit).

DETAILED DESCRIPTION:
The long term goal of the investigators work is to implement real world CPR training strategies that match training locales with at-risk populations, maximize resuscitation skill retention, and promote willingness to act. To accomplish this, the investigators will empower stakeholders at UPHS and local area hospitals to develop local implementation approaches, using either volunteers or nursing staff as training proctors. These stakeholders will be studied as a research subset. The training proctors will train family members or friends of patients at risk for cardiac arrest using either a video-only method or video self-instruction (VSI) kit, and empower them with the lifesaving skill of CPR. The investigators will use the American Heart Association's CPR Anytime VSI kit which comes equip with a DVD and inflatable manikin. For the group receiving the video-only method, the investigators will remove the inflatable manikin and train the subjects with the DVD. The investigators will randomize family members of high risk for CA to either the video-only or VSI kit method of training. The training proctors will be instructed to switch training methods every 6 months. The investigators will follow up with the study subjects and conduct CPR skills tests from 6 to 12 months from time of training to assess whether the subjects retained their skills or if they had an opportunity to use the skills that they learned. The investigators will also gather information on how the subjects would like to be encouraged to practice their skills. The investigators will send a reminder notification every two months following training, to encourage the subjects to refresh their training skills. At the follow-up skills test at 6 to 12 months, we will administer a survey to assess whether the prompting encouraged the subjects to practice their skills.

ELIGIBILITY:
Inclusion Criteria:

* Family Members of Patients with known coronary disease or cardiovascular risk factors, such as history of diabetes and hypertension.

Exclusion Criteria:

* If someone is physically unable to undergo CPR Training

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1870 (Actual)
Dates: Start 2011-11; Primary Completion 2015-07 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
CPR Skills Performance and Retention | 6 months
  To assess skills performance and retention by trainees (family members and friends) taught using a video-only method or video self-instruction kit. To assess whether prompting or reminding subjects (family members and friends) might encourage the subjects to practice their CPR skills and improve skills at time of testing. Subjects skills will be tested at 6 and 12 months period of time.

SECONDARY OUTCOMES:
Assessing CPR Training Proctors (Nurses or Volunteers) | At 3 months, 6 months, 9 months and 12 months
  To determine if volunteers or nursing staff can adequately implement a CPR training program to "at risk" family members or friends of patients hospitalized for cardiac risk factors. Subjects will be surveyed every 3 months to assess feasibility.
Assess prompting to encourage CPR skills retention | up to 1 year
  To assess whether prompting subjects every two months encourages them to practice and retain the skills that they learned.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin S. Abella, MD, MPhil, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blewer AL, Leary M, Decker CS, Andersen JC, Fredericks AC, Bobrow BJ, Abella BS. Cardiopulmonary resuscitation training of family members before hospital discharge using video self-instruction: a feasibility trial. J Hosp Med. 2011 Sep;6(7):428-32. doi: 10.1002/jhm.847. Epub 2010 Nov 8. PMID 21916007
- [Background] Blewer AL, Leary M, Esposito EC, Gonzalez M, Riegel B, Bobrow BJ, Abella BS. Continuous chest compression cardiopulmonary resuscitation training promotes rescuer self-confidence and increased secondary training: a hospital-based randomized controlled trial*. Crit Care Med. 2012 Mar;40(3):787-92. doi: 10.1097/CCM.0b013e318236f2ca. PMID 22080629
- [Derived] Blewer AL, Putt ME, Becker LB, Riegel BJ, Li J, Leary M, Shea JA, Kirkpatrick JN, Berg RA, Nadkarni VM, Groeneveld PW, Abella BS; CHIP Study Group*. Video-Only Cardiopulmonary Resuscitation Education for High-Risk Families Before Hospital Discharge: A Multicenter Pragmatic Trial. Circ Cardiovasc Qual Outcomes. 2016 Nov;9(6):740-748. doi: 10.1161/CIRCOUTCOMES.116.002493. Epub 2016 Oct 4. PMID 27703033